CLINICAL TRIAL: NCT00135018
Title: Phase II Study on the Neoadjuvant Use of Chemotherapy and Celecoxib Therapy in Patients With Invasive Breast Cancer
Brief Title: Study on the Neoadjuvant Use of Chemotherapy and Celecoxib Therapy in Patients With Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organisation for Oncology and Translational Research (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEC-DOC-CXB-A3
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib and chemotherapy

SUMMARY:
This study will investigate whether cyclooxygenase inhibition with celecoxib will add any benefit to preoperative chemotherapy alone for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be free of psychiatric or addictive disorders and mentally able to follow prescription instructions and able to give written informed consent. The patient must consent to be in the study and must sign an approved consent form conforming to institutional guidelines.
* The patient must be aged 18 years or older.
* The diagnosis of invasive adenocarcinoma of the breast must be confirmed by core or Tru-cut biopsy and the interval between initial histological diagnosis of breast cancer and registration must not be more than 1 month.
* The primary tumor within the breast must be palpable and measurable on clinical examination and ultrasound, and must be confined to one breast. For patients with clinically negative axillary nodes, the primary tumor size must be between 2 to 7 cm. For patients with clinically positive axillary nodes, any primary tumor size up to 7 cm is acceptable (T2-3, N0, M0 or T1-3, N1, M0).
* ECOG performance status of 0-1 or a corresponding Karnofsky performance status of at least 70.
* Within one month prior to the time of registration, the patient must have had the following: history, physical examination, blood tests, tumor estrogen and progesterone receptor status assessment, chest X-ray, bone scan, abdominal ultrasound, bilateral mammogram, and electrocardiogram (ECG).
* Hematology parameters: white blood cell (WBC) at least 2500/mm3; neutrophil count at least 2,000/mm3; platelet count at least 100,000/mm3; and hemoglobin at least 10g/dL. Other laboratory parameters: total serum bilirubin not exceeding 2 times institutional upper limit of normal (ULN); AST not exceeding 2 times ULN; ALT not exceeding 2 times ULN; alkaline phosphatase not exceeding 2 times ULN; and serum creatinine not exceeding 2 times ULN. In borderline cases, inclusion into the study is left to the judgment of the principal investigator.
* The patient must have adequate ventricular function with left ventricular ejection fraction (LVEF) not less than 55% by echocardiogram scan.
* Patients with prior non-breast malignancies are eligible if they have been disease free for more than 5 years and if they have not received any chemotherapy, immunotherapy, hormonal therapy or radiation therapy within the last 5 years. Patients with curatively treated non-melanoma skin cancer and carcinoma in situ of the cervix are eligible even if diagnosed within the last 5 years prior to registration.
* Patients receiving any sex hormonal therapy e.g., birth control pills, ovarian hormonal replacement therapy, etc., are eligible if such therapy is discontinued 1 month prior to registration.

Exclusion Criteria:

* Male patients
* Patients with distant metastasis, including skin involvement beyond the breast area. Patients with ulceration, erythema and infiltration of the skin (complete fixation), inflammatory breast cancer or peau d'orange (edema) of any magnitude. (Tethering or dimpling of the skin or nipple inversion should not be interpreted as skin infiltration and patients with these conditions are eligible.)
* Patients with ipsilateral lymph nodes that are clinically fixed to one another or to other structures (N2 disease).
* Patients with a mass in the opposite breast, which is suspicious for malignancy, unless there is biopsy proof that the mass is not malignant.
* Patients with multiple, bilateral breast cancer or suspicious palpable nodes in the contralateral axilla or patients with palpable supraclavicular or infraclavicular nodes, unless there is biopsy proof that the nodes are not involved with malignancy.
* Postmenopausal patients with both positive estrogen and progesterone receptor status and negative lymph node involvement.
* Pregnant women or women with suspected pregnancy at the time of registration and lactating women are not eligible for the study.
* Patients with prior history of invasive breast cancer; patients with ipsilateral new cancer/recurrence after treatment of in-situ breast cancer; or patients who have received prior therapy for breast cancer, including chemotherapy, immunotherapy, hormonal therapy or radiation therapy.
* Patients who have received any prior anthracycline or docetaxel therapy for any malignancy.
* Patients with serious cardiac illness or medical conditions including, but not confined to:

  * History of documented congestive heart failure (CHF);
  * High-risk uncontrolled arrhythmias;
  * Angina pectoris requiring antianginal medication;
  * Clinically significant valvular heart disease;
  * Evidence of transmural infarction on ECG; or
  * Poorly controlled hypertension (e.g. systolic > 180mmHg or diastolic greater than 100mmHg).
* Patients with any abnormalities in the ECG, e.g., ventricular hypertrophy, even if they demonstrate adequate ventricular function by echocardiogram.
* Patients with active or chronic documented infection at the time of registration.
* Patients with pre-existing peripheral neuropathy (grade 2 or greater according to National Cancer Institute Adverse Event [NCI AE] v 3.0) and patients under risk of developing peripheral neuropathy, i.e., poorly controlled diabetes mellitus.
* Patients with rheumatic disease and patients under cyclooxygenase-2 inhibitor medication.
* Patients who are hepatitis B and/or hepatitis C carriers.
* Patients with known hypersensitivity or contraindication to any study or pre- medications or products formulated in polysorbate 80.
* Patients judged by the investigator to be unfit to be enrolled into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-02; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis WC Chow, Principal Investigator — UNIMED Medical Institute
Locations (1):
- UNIMED Medical Institute, Hong Kong, Hong Kong